CLINICAL TRIAL: NCT04095923
Title: A Social Media Game to Increase Physical Activity Among Older Adult Women
Acronym: CHALLENGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute on Aging (NIA) (NIH); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-0158; R01AG064092 (NIH)
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Aging
Keywords: Physical activity; Social media; Wearable; Intrinsic motivation; Game; Women's health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social media game (Experimental): Private Facebook group with weekly walking challenges, Fitbit wearable activity monitor, and brief counseling
  Interventions: Behavioral: Social media game
- Standard self-regulation (Active Comparator): Fitbit wearable activity monitor and brief counseling
  Interventions: Behavioral: Standard self-regulation

INTERVENTIONS:
Behavioral: Social media game — Participants will engage in weekly challenges that require them to take photographs of interesting things they discover during their walks. They will post and discuss these photographs with other participants on a private social media page. They will track their steps using a wearable activity monitor and receive brief standard self-regulatory counseling.
  Arms: Social media game
Behavioral: Standard self-regulation — Participants will track their steps using a wearable activity monitor and receive brief standard self-regulatory counseling.
  Arms: Standard self-regulation

SUMMARY:
This study will test the effects of a social media game on the physical activity of older adult women. The game will consist of playful weekly challenges that require sharing photographs on a private social media group and also wearing an activity monitor to track steps. Participants will be randomized to this game group or to receive the activity monitor only.

DETAILED DESCRIPTION:
Older adult women are at risk for negative health impacts of physical inactivity, but current strategies to increase their activity have had disappointing long-term results. The intervention tested in this study seeks to test an innovative intervention that targets older womens' perceptions of enjoyment and their personal identity and values. The investigators will test the efficacy of a 12-month social media-based physical activity intervention for sedentary older adult women. Participants will be randomized to receive a standard Fitbit-only intervention or to an enhanced Fitbit + weekly social challenges intervention. The investigators hypothesize that participants in the enhanced intervention will demonstrate greater increases in autonomous regulation and objectively-measured steps as compared to those in the standard intervention. The investigators will also measure outcomes after a 6 month maintenance period (18 months after beginning the intervention). Additional outcomes will include engagement with the social network and self-reported playful experiences.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age between 65 and 85
3. Able to read and understand English
4. Willingness to be randomized to any condition
5. Daily availability of an iOS or Android mobile device that is capable of taking and sending photos
6. Willingness to use a private Facebook group
7. Sufficient internet access to post photos to Facebook at least once per week
8. Having an existing Facebook account or willingness to create one

Exclusion Criteria:

1. Unable to find transportation to the study location
2. Unable to walk for exercise (self-report)
3. Walk <475 meters in 6 minute walk test during baseline assessment
4. Stroke, hip fracture, hip or knee replacement, or spinal surgery in the past 6 months
5. Participant answered "yes" to any question on the PAR-Q+ and does not provide a doctor's note giving permission to begin a physical activity program
6. Self-reported weekly PA ≥ 150 minutes
7. BMI under 18 or over 40
8. Participant reports psychological issues that would interfere with study completion. Examples will be provided to illustrate potential psychological issues, such as dementia or schizophrenia.
9. Participant plans to move away from the Galveston-Houston area or to be out of town for more than 2 weeks at a time during the study period
10. Clinical judgment concerning safety
11. Currently participating in an organized commercial or research physical activity program
12. Uses a wearable activity monitor other than a simple pedometer and is unwilling to stop during the trial
13. Another member of the household is a participant or staff member on this trial

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Participants must self-report as women
Enrollment: 300 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Walking physical activity as measured by daily steps at 12 months | Baseline to 12 months
  Mean of daily steps taken from accelerometers worn for a 7 day period

SECONDARY OUTCOMES:
Walking physical activity as measured by daily steps at 6 months | Baseline to 6 months
  Mean of daily steps taken from accelerometers worn for a 7 day period
Walking physical activity as measured by daily steps at 18 months | Baseline to 18 months
  Mean of daily steps taken from accelerometers worn for a 7 day period
Intrinsic regulation | Baseline to 6 months
  Self-reported intrinsic regulation on a scale from 0 (least motivated) to 4 (most motivated) using the Behavioral Regulation in Exercise Questionnaire - 3
Integrated regulation | Baseline to 6 months
  Self-reported integrated regulation on a scale from 0 (least motivated) to 4 (most motivated) using the Behavioral Regulation in Exercise Questionnaire - 3
Autonomous regulation | Baseline to 6 months
  Composite of subscales for intrinsic, integrated, and identified regulation as measured on a scale from 0 (least motivated) to 4 (most motivated) using the Behavioral Regulation in Exercise Questionnaire - 3
Basic psychological needs | Baseline to 6 months
  Perceptions of autonomy, competence, and relatedness on a scale from 1 (don't agree) to 5 (completely agree) using the Psychological Needs in Exercise Scale
Physical activity as measured by minutes of moderate-vigorous intensity physical activity at 6 months | Baseline to 6 months
  Mean daily minutes of moderate-vigorous intensity physical activity taken from accelerometers for a 7 day period
Physical activity as measured by minutes of moderate-vigorous intensity physical activity at 12 months | Baseline to 12 months
  Mean daily minutes of moderate-vigorous intensity physical activity taken from accelerometers for a 7 day period
Physical activity as measured by minutes of moderate-vigorous intensity physical activity at 18 months | Baseline to 18 months
  Mean daily minutes of moderate-vigorous intensity physical activity taken from accelerometers for a 7 day period

OTHER OUTCOMES:
Exercise identity | Baseline to 6 months
  Perceptions of exercise identity on a scale from 1 (strongly disagree) to 7 (strongly agree) on the Exercise Identity Scale
Engaged living | Baseline to 6 months
  Perceptions of value-based living on a scale of 1 (completely disagree) to 5 (completely agree) on the Engaged Living Questionnaire
Playful experiences | Baseline to 6 months
  Self-reported playful experiences during play of the game on a scale of 1 (totally disagree) to 5 (totally agree) using the Playful Experiences Questionnaire
Usability | Baseline to 6 months
  Self-reported usability of the social media group on a scale of 1 (strongly disagree) to 5 (strongly agree) using the System Usability Scale
Acceptability of walking challenge game | Baseline to 6 months
  Self-reported acceptability of challenges on a scale of 1 (strongly disagree) to 5 (strongly agree)
Engagement in the social media group | Baseline to 12 months
  Objectively measured number of posts, comments, and reactions in the Facebook group
Days the activity monitor was worn | Baseline to 12 months
  Objectively measured days the wearable activity monitor was worn during the intervention period
Enjoyment of each weekly challenge | Baseline to 12 months
  Self-reported enjoyment measured via weekly text message inquiring as to enjoyment on a scale from 1 (strongly disagree) to 7 (strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lyons, PhD, MPH, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will provide access to all data, regardless of publication, collected as a part of this project. All external investigators must submit a written request identifying their research question(s) and specifying the data they would like to analyze. The request must include a data security plan and explanation of how the data will be stored and who will have access. All requests will be reviewed by the investigators in conjunction with UTMB's Institute for Translational Sciences key resources (in particular, the regulatory and ethics resources) to be sure appropriate NIH requirements are followed.
Supporting Information: Study Protocol, SAP
Time Frame: Data will only be available upon request
Access Criteria: All external investigators must submit a written request identifying their research question(s) and specifying the data they would like to analyze. The request must include a data security plan and explanation of how the data will be stored and who will have access. All requests will be reviewed by the investigators in conjunction with UTMB's Institute for Translational Sciences key resources (in particular, the regulatory and ethics resources) to be sure appropriate NIH requirements are followed.

REFERENCES:
- [Derived] Robertson MC, Swartz MC, Basen-Engquist KM, Li Y, Jennings K, Thompson D, Baranowski T, Volpi E, Lyons EJ. A social media game to increase physical activity among older adult women: protocol of a randomized controlled trial to evaluate CHALLENGE. BMC Public Health. 2024 Aug 12;24(1):2172. doi: 10.1186/s12889-024-19662-9. PMID 39135010